CLINICAL TRIAL: NCT06885697
Title: Phase 1 Study With Dose Expansion of the Anti-Mesothelin TNaive/SCM hYP218 (TNhYP218) CAR T Cells in Participants With Mesothelin-Expressing Solid Tumors Including Mesothelioma
Brief Title: Anti-Mesothelin TNaive/SCM hYP218 (TNhYP218) CAR T Cells in Participants With Mesothelin-Expressing Solid Tumors Including Mesothelioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10002021; 002021-C
Record Dates: First submitted 2025-03-19; First posted 2025-03-20 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12-17

CONDITIONS: Mesothelioma; Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Thymus Neoplasms; Colonic Neoplasms
Keywords: Peritoneal Mesothelioma; Thymic Carcinoma; Colon Cancer; Gastric Cancer; Lung Cancer; Ovarian Cancer; Pancreatic Cancer; mesothelin expressing solid tumors; CAR T cell therapy; Gene Therapy
MeSH Terms: conditions — Mesothelioma; Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Thymus Neoplasms; Colonic Neoplasms; Thymoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- 1/Dose Escalation (Experimental): Participants with mesothelin expressing tumors will undergo lymphodepletion and will receive TNhYP218 CAR T cells at escalating doses
  Interventions: Device: mesothelin expression testing; Biological: TNhYP217 CAR T Cells; Drug: fludarabine; Drug: cyclophosphamide
- 2/Dose Expansion (Experimental): Participants with mesothelioma will undergo lymphodepletion and will receive TNhYP218 CAR T cells at the RP2D determined in Arm 1
  Interventions: Device: mesothelin expression testing; Biological: TNhYP217 CAR T Cells; Drug: fludarabine; Drug: cyclophosphamide

INTERVENTIONS:
Device: mesothelin expression testing — Assay done at screening to determine mesothelin expression levels
Biological: TNhYP217 CAR T Cells — Variable doses, administered intravenously on Day 0
Drug: fludarabine — 30 mg/m^2 IV infusion administered followed by cyclophosphamide on days both are given. Daily x 4 doses on Day -7, -6, -5 and -4
Drug: cyclophosphamide — 600 mg/m^2 IV infusion. Daily x 3 doses on Day -6, -5, -4

SUMMARY:
Background:

Mesothelioma is an aggressive cancer that grows in the linings of the body; this can include the membranes that line the heart, lungs, and internal organs. Mesothelin (MSLN) is a protein that appears in high numbers in many tumors, including mesothelioma. Researchers are developing a new treatment that collects a person s own immune cells (T cells); the T cells are genetically modified to target and kill tumor cells with high levels of MSLN.

Objective:

To test a new treatment (TNhYP218 CAR T cells) in people with solid tumors including mesothelioma.

Eligibility:

People aged 18 and older with solid tumors including mesothelioma that returned or spread after standard treatment.

Design:

Participants will be screened. A small piece of tissue will be cut from a tumor (biopsy). The sample will be tested to see if it has enough MSLN.

Participants will undergo leukapheresis: Blood will be taken from their body through a vein. The blood will pass through a machine that separates out the T cells. The remaining blood will be returned to the body through a different vein.

Participant s T cells will be modified in a lab to produce TNhYP218 CAR T cells.

Participants will enter the hospital. For 7 days, they will receive drugs to prepare their bodies for the study treatment.

TNhYP218 CAR T cells will be administered into a vein. Participants will remain in the hospital for at least 7 more days.

After discharge, participants will have follow-up visits for 5 years. These visits may include imaging scans, blood and heart tests, and a new biopsy.

Long-term follow-up will continue another 10 years.

DETAILED DESCRIPTION:
Background:

* Mesothelin (MSLN), a cell surface glycoprotein, normally expressed on the mesothelial cells lining the pleura, peritoneum, and pericardium, is highly expressed in many cancers including mesothelioma, ovarian, lung, thymic, colorectal, pancreatic, and gastric cancers, making it an attractive target for immunotherapy.
* Adoptive cell therapy using CAR T cells exploits the ability of these modified T cells to recognize and kill their target. Several mesothelin directed CAR T cell therapies have been evaluated in clinical trials, but thus far have not resulted in significant anti-tumor efficacy.
* Many antibodies used to make anti-mesothelin CAR T cells bind to the immunogenic distal region of mesothelin, away from the cell membrane.
* hYP218 CAR T cells target membrane-proximal region of mesothelin and in pre-clinical studies have shown increased tumor killing and persistence compared to CAR T cells binding to membrane distal region of mesothelin.
* Naive/SCM T cells have stem cell like properties and have increased persistence and decreased exhaustion in tumors.
* We hypothesize that TNaive/SCM anti-mesothelin, TNhYP218 CAR T cells will have enhanced anti-tumor activity and increased persistence in participants with mesothelioma and other mesothelin expressing cancers.

Objectives:

* Part 1- Dose escalation: Establish the recommended phase 2 dose (RP2D) of TNhYP218 CAR T cells based on dose-limiting toxicity (DLT) of defined adverse events (AEs).
* Part 2- Dose expansion: Determine the preliminary objective response rate of TNhYP218 CAR T cells in a limited number of participants with mesothelioma treated at the RP2D.

Eligibility:

* Age 18 or older
* Must have unresectable, histologically confirmed, recurrent, locally advanced, or metastatic mesothelioma, and other mesothelin expressing solid tumors.
* Tumor must be positive for mesothelin in more than half of the cancer cells.
* Participants must have an ECOG performance status of 0 or 1.
* Participants must have adequate organ function.

Design:

* Phase 1 dose-escalation study of TNhYP218 CAR T cells, with a small expansion cohort.
* Participants will undergo leukapheresis for cell manufacture, followed by lymphodepletion with chemotherapeutic drugs, followed by infusion of TNhYP218 CAR T cells.
* Participants will be followed for safety for up to 15 years per FDA requirement.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria. For this protocol, treatment initiation is defined as the first day of lymphodepleting chemotherapy.

* Participant must have unresectable, locally advanced, or metastatic, or recurrent mesothelioma and other mesothelin expressing solid tumors. For participants with mesothelioma only those with epithelioid or biphasic histology (with >80% epithelioid component) will be eligible. The diagnosis will be confirmed by the Laboratory of Pathology, CCR, NCI.
* Participant must have progressed on at least one FDA-approved systemic therapy considered standard of care for their tumor type. There is no limit on the number of prior treatment regimens. Note: Given the aggressive nature of pancreatic cancer, otherwise eligible individuals with this cancer type can undergo leukapheresis before or while they are getting their frontline treatment as long as they meet all other inclusion criteria. However, TNhYP218 CAR T cells will only be administered after progression on first line standard of care therapy.
* Participant must have at least 1 measurable lesion by RECIST version 1.1.
* Tumor must have MSLN positivity of 2+ to 3+ in >= 50% cancer cells by immunohistochemistry on freshly collected biopsy or archival tissue.
* Age >= 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants must have adequate organ and marrow function as defined below:

System: Laboratory Value

Hematological

* Hemoglobi: >=9 g/dL(a)
* absolute neutrophil count: >=1,500/mcL
* platelets: >=100,000/mcL

Hepatic

* total bilirubin: <=2.5 X institutional ULN OR direct bilirubin ULN for participants with total bilirubin levels >1.5 X ULN
* AST and ALT <= 2.5 X institutional ULN (<= 5 X ULN for participants with liver metastases)

Renal

* Creatinine OR: <=1.5 X ULN OR
* Calculated(b) creatinine clearance (GFR can also be used in place of creatinine or CrCl) >= 50 mL/min for participant with creatinine levels > 1.5 X institutional ULN

Coagulation

* International normalized ratio (INR) OR prothrombin time (PT): <=1.5 X ULN unless participant is receiving anticoagulant therapy if PT or aPTT is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT): <=1.5 X ULN unless participant is receiving anticoagulant therapy if PT or aPTT is within therapeutic range of intended use of anticoagulants

ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.

1. Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
2. Creatinine clearance (CrCl) should be calculated per institutional standard.

   * Normal cardiac ejection fraction (>= 45% by echocardiogram) and no evidence of hemodynamically significant pericardial effusion as determined by an echocardiogram.
   * Room air oxygen saturation of 90% or greater.
   * Treatment-related toxicities from prior treatments must be resolved to <= grade 2.
   * Participants with CNS metastases, leptomeningeal disease or carcinomatous meningitis are eligible if they are asymptomatic, have completed their treatment for CNS disease and have recovered from the acute effects of radiation therapy or surgery prior to study entry. Participants must have radiographically stable CNS disease without associated edema at least three months prior to study entry. Additionally, participants have had to have discontinued corticosteroid treatment or non-prophylactic antiseizure medications for these metastases at least four weeks prior to study entry.
   * Participants of child-bearing potential and participants who can father children must agree to use highly effective contraception or abstinence.
   * Participants who are nursing or plan to nurse a child must agree to discontinue/postpone nursing for the duration of study therapy and for 12 months after the administration of the cell product or for 4 months from the time no evidence of persistence/gene modified cells is documented in the participant s blood.
   * Ability of participant to understand and the willingness to sign a written informed consent document.

   EXCLUSION CRITERIA:

   An individual who meets any of the following criteria will be excluded from participation in this study:
   * Prior systemic therapy, an investigational therapy, radiation, and/or surgery within 14 days prior to leukapheresis and 21 days prior to lymphodepleting chemotherapy.
   * Prior administration of anti-PD-1 or anti-PD-L1 antibodies or other agents that in the opinion of the PI can stimulate immune activity and interfere with an infusion of CAR-T cells within 8 weeks prior to treatment initiation.
   * Participants with any form of primary immunodeficiency (e.g. severe combined immunodeficiency).
   * Participants with active or history of autoimmune or immune mediated disease such as multiple sclerosis, lupus, inflammatory bowel disease, rheumatoid arthritis, or small vessel vasculitis. NOTE: Participants with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible.
   * History of severe immediate hypersensitivity reaction to cyclophosphamide or fludarabine.
   * Therapeutic doses of systemic corticosteroid therapy within 14 days prior to treatment initiation. Physiological doses of steroids (up to 5mg/day of prednisolone or equivalent) are allowed. Corticosteroid creams, ointments, and eye drops are allowed.
   * Participants with lung fibrosis, inflammatory lung disease or evidence of pneumonitis on baseline imaging studies or medical history of these disorders.
   * Participant has any other prior or concurrent malignancy with the following exceptions:

     * Adequately treated basal cell or squamous cell carcinoma
     * In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 12 months prior to initiation of study therapy.
     * Treated non-melanoma skin cancer.
     * Stage 0 or 1 melanoma completely resected at least 12 months prior to initiation of study therapy.
     * Successfully treated organ-confined prostate cancer with no evidence of progressive disease based on PSA levels and are not on active therapy.
     * A primary malignancy which has been completely resected and in complete remission for >= 5 years.
   * Electrocardiogram showing a QTc interval > 450 msec in males and > 470 msec in females (> 80 msec for participants with bundle branch block). Either Fridericia s or Bazett s formula may be used to correct the QT interval.
   * Participant has active infection with HIV, hepatitis B virus, HCV, or HTLV as defined below:

     * Positive serology for HIV, HTLV-1, or HTLV-2.
     * Active hepatitis B infection as demonstrated by test for hepatitis B surface antigen. Participants who are hepatitis B surface antigen negative but are hepatitis B core antibody positive must have undetectable hepatitis B DNA and receive prophylaxis against viral reactivation.
     * Active hepatitis C infection as demonstrated by hepatitis C RNA test. Participants who are HCV antibody positive will be screened for HCV RNA by any reverse transcription PCR or branched DNA assay. If HCV antibody is positive, eligibility will be determined based on a negative screening RNA value.
   * Participant is pregnant or intends to be pregnant during the required period of contraception for participants of childbearing potential.
   * Participants who received live or attenuated vaccine or virus-based vaccine within 30 days before initiation of treatment initiation
   * Participants with a history of seizure disorder unless due to now treated metastatic lesions.
   * Ongoing uncontrolled intercurrent illness, including but not limited to ongoing or active infection, that would impact participant safety or limit compliance with study requirements.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2034-06-01 (Estimated); Study Completion 2044-06-01 (Estimated)

PRIMARY OUTCOMES:
Establish the recommended phase 2 dose (RP2D) of TNhYP218 CAR T cells based on dose-limiting toxicity (DLT) of defined adverse events (AEs). | DLT assessment will occur in participants in the dose escalation cohort daily on days 0-4, on day 7, on day 21 and during week 4.
  The highest dose level below the maximum administered dose at which no more than 1 of 6 participants experience DLT from the initiation of CAR-T cell infusion (day 0) through day 28 after infusion (day 28).
Determine the preliminary objective response rate of TNhYP218 CAR T cells in a limited number of participants with mesothelioma treated at the recommended phase 2 dose. | assessed based on imaging studies at weeks 4, 8, 12 then every 12 weeks through disease progression or week 108, whichever occurs first.
  The proportion of mesothelioma participants with partial response or complete response at the recommended phase 2 dose.

SECONDARY OUTCOMES:
Near term safety of autologous genetically modified TNhYP218 CAR T cells in adult study participants with mesothelin expressing unresectable, metastatic, or recurrent mesothelioma and other mesothelin expressing solid tumors. | Assessments will occur daily during lymphodepletion, on day of cell infusion (D0), D10, D21, every 2 weeks from W4 to W8, then every 4 weeks through W 24 or disease progression.
  The near-term safety of the study therapy will be evaluated by reporting the grade and type of toxicity at each dose level.
Long term safety of autologous genetically modified TNhYP218 CAR T cells in adult study participants with mesothelin expressing unresectable, metastatic, or recurrent mesothelioma and other mesothelin expressing solid tumors. | Monitored at baseline, weeks 4, 12, 24 and 48 after cell infusion and annually thereafter for up to 15 years if positive during year 1 or warranted based on clinical history collected annually during15 year follow-up.
  The long-term safety will be assessed by the presence of RCL as well as clinical assessments.
Determine the objective response rate of TNhYP218 CAR T cells in participants with mesothelin expressing solid tumors treated at doses other than the RP2D | assessed based on imaging studies at weeks 4, 8, 12 then every 12 weeks through disease progression or week 108, whichever occurs first.
  The proportion of participants with partial response or complete response at doses other than the recommended phase 2 dose.
Determine progression free survival in participants with mesothelin expressing solid tumors | Assessed based on imaging studies at weeks 4, 8, 12 then every 12 weeks through disease progression or week 108, whichever occurs first.
  The duration of time from start of treatment (lymphodepletion) to time of progression or death, whichever occurs first.
Determine duration of response in participants with mesothelin expressing solid tumors | Assessed based on imaging studies at weeks 4, 8, 12 then every 12 weeks through disease progression or week 108, whichever occurs first.
  The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Determine overall survival in participants with mesothelin expressing solid tumors | Assessed from physical exams performed on D10, D21, W4, W6, W8, then every 4 weeks through W 24, and with semiannual remote assessments following active follow up through year 5.
  The duration of time from start of treatment (lymphodepletion) to time of death from any cause.
Evaluate feasibility of manufacturing TNhYP218 CAR T cells from participants with mesothelin expressing solid tumors. | Assessed prior to cell infusion (Day 0).
  The fraction of participants with cell products produced with Tna(SqrRoot) ve/scm cells
Assess the tolerability of lymphodepletion followed by TNhYP218 CAR T-cell infusion in participants with mesothelin expressing solid tumors | Assessed through cell infusion (Day 0)
  -The fraction of participants able to receive all protocol therapy without treatment delay.-The fraction of participants able to receive cell product without interruption due to infusion related reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Raffit Hassan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Management and Sharing (DMS) Policy, which applies to all new and ongoing NIH-funded research in the IRP, as of January 25, 2023, that is associated with a ZIA, with a clinical protocol that undergoes scientific review and/or will involve genomic data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available as soon as possible or at the time of associated publication. Data not published in a manuscript will be shared via public source once the data set completes QC.
Access Criteria: The scientific data will be findable by key words or MeSH terms used during publication of manuscripts.@@@@@@All scRNA seq data will be uploaded to dbGaP and accession numbers will be shared.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_002021-C.html